CLINICAL TRIAL: NCT07278167
Title: Analysis of Risk Factors and Predictive Value for 28-Day Mortality in Patients With Sepsis and Nutritional Risk
Brief Title: Analysis of Risk Factors and Prognostic Predictive Value in Sepsis Patients With Nutritional Risk
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Inner Mongolia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AHInnerMongolia-NT
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Nutritional Risk
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- survivors/non-survivors
  Interventions: Other: Retrospective data analysis, no intervention

INTERVENTIONS:
Other: Retrospective data analysis, no intervention — Retrospective data analysis, no intervention

SUMMARY:
Sepsis is a common critical illness in intensive care units, characterized by systemic inflammatory response, immune dysfunction, microcirculatory issues, and multi-organ failure. These factors lead to high mortality rates and poor prognoses for patients. Nutritional risk is a significant complication in patients with sepsis, with a prevalence of 38% - 78. Sepsis-induced hypermetabolism and hypercatabolism result in increased energy expenditure and accelerated protein breakdown in affected patients, which subsequently exacerbates the risk of malnutrition. Malnutrition weakens immune function, reduces resistance to infections, and impairs immune regulation in sepsis patients. It worsens organ dysfunction, prolongs ICU hospitalization, and increases morbidity and mortality rates. Early identification and intervention for potential risk factors in patients with sepsis, particularly those with nutritional risk, is crucial for enhancing their prognosis. There is a notable lack of sensitive indicators for assessing the prognosis of sepsis patients at nutritional risk. Recent studies have begun exploring physical assessment measures in ICU settings as accessible and noninvasive tools for evaluation. This study aims to investigate the predictive value of nutritional laboratory indicators and physical measurements regarding the 28-day outcomes of ICU patients with sepsis and nutritional risk, providing a foundation for early clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Met the diagnostic criteria for sepsis 3.0
2. Met the diagnostic criteria for nutritional risk (NRS-2002 score ≥ 3)
3. ICU stay≥2 days
4. Age ≥ 18

Exclusion Criteria:

1. Edema
2. Tumor patients
3. Pregnancy
4. Lack of complete laboratory results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sepsis with nutritional risk
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
28-day clinical outcome | 28day

CONTACTS AND LOCATIONS:
Locations (1):
- Jing Lin, Hohhot, China

IPD SHARING:
Plan to Share IPD: Undecided